CLINICAL TRIAL: NCT03994562
Title: Determinants of Frailty Among of Informal Caregivers of Demented Patient Evaluated in Day Care Hospital.
Brief Title: Determinants of Frailty Among of Informal Caregivers of Demented Patient
Acronym: DELFAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02925-50
Record Dates: First submitted 2019-01-22; First posted 2019-06-21 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Fragility
Keywords: Frailty; Caregivers; Zarit scale
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty, a transitional state between successful and pathological aging, may be benefit from early multi-interventional intervention. Fried's criteria are the more commonly used criteria to diagnose frailty. The caregivers' burden increases caregivers' morbidity .The main objective of the study was to assess the relationship between frailty among informal caregivers of demented patients and the caregiver's burden (Zarit scale). The Secondary objective was to assess determinants of frailty among caregivers.

DETAILED DESCRIPTION:
Frailty, a transitional state between successful and pathological aging, may be benefit from early multi-interventional intervention.

Fried's criteria are the more commonly used criteria to diagnose frailty :

* Loss of weight > 4.5 kg over one year,
* Self-reported exhaustion,
* Low muscle strength (handgrip <20% norm for age and sex),
* Low physical activity
* Low gait speed (<0.8m/s). According to the number of Fried's criteria, subjects are considered frail (≥ 3 Fried's criteria), pre-frail (1-2 Fried's criteria) or robust (0 Fried's criterion).

A large proportion of care is believed to be delivered by informal caregivers (e.g., spouses, next of kin). The caregivers' burden experienced as "enduring stress and frustration" due to caregiving, affects caregivers' mental health with depression, anxiety and sleep disorders, increases caregivers' morbidity and mortality. Multi-interventional studies (including physical and psychological wellbeing) have proven their accuracy to improve quality of life of caregivers.

In France, caregivers (>60 years) of demented people number have been estimate to 3.3 million (DREES).

For more than one year, in the Broca memory center (3000 patients/ years), caregivers can benefit from a comprehensive medico-psychosocial assessment during a day care hospital. Frailty is assessed in usual care. Two caregivers a week benefit from this assessment. The same day care hospital has been implemented in the "Paul Brousse" hospital (100 patients/year) : One caregiver a week benefit from this assessment.

Main objective:

To assess the relationship between frailty among informal caregivers of demented patients and the caregiver's burden (Zarit scale).

Secondary objective:

To assess determinants of frailty among caregivers.

Main outcome :

Caregiver burden will be determined according to the Zarit scale. The Zarit scale is an auto-questionnaire which includes 22 questions (rated from 0 to 4 points) and scores out of 88. A higher score reflects a higher caregiver burden.

Frailty will be defined by Fried criteria. Subjects will be considered as frail (≥ 3 Fried's criteria), pre-frail (1-2 Fried's criteria) or robust (0 Fried's criteria).

Secondary outcomes

* Age, sex, educational level
* Treatments et polypharmacy (≥ 4 treatments)
* Neuropsychological test if cognitive complaint : caregivers will be categorized as cognitively normal, mild cognitive impairment or dementia.
* Depression according to the Pichot scale and the Geriatric Depression Scale.
* Anxiety according to the Goldberg scale
* Nutritional Assessment: mini nutritional assessment and body mass index.

Feasibility :

Eighty caregivers will be included in the Broca hospital and 40 in the Paul Brousse hospital. To reach the calculated number of subjects to include (n=120), inclusions will take place during 1 year and a half.

Statistical analysis

Main objective :

To disclose a difference in the Zarit score of 11 points (retrospective analysis of collected data) with 80% power and α 5% risk, 120 subjects have to be included. The population will be described and factors associated with the Zarit scale in uni-variate analysis will be studied in a multiple linear regression model.

Analysis will be also performed according to 3 groups: frail, pre-frail and robust.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of demented patients ,
* over > 65 years old,
* who accept exhaustive evalutaion in day care hospital, who agree for ther data to be recorded (anonymously) for an observational study

Exclusion Criteria:

* No affliation to French social insurance system
* People under tutorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: caregivers of demented patients who are aware of the day care hospital and who want to be assesed
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the emotional, physical and financial burden on a caregiver according Zarit burden scale | Day 0

SECONDARY OUTCOMES:
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) scores | Day 0
Screening for a nutritional disorder according Body Mass Index (BMI) score | Day 0
Assessment of verbal episodic memory according Grober and Buschke's test | Day 0
Screening of the undernutrition according mini nutritional assessment (MNA) | Day 0
Assessment of anxiety according Goldberg scale | Day 0
Assessment of humor in geriatrics according Geriatric Depression Scale (GDS) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Duron, Md, PHd, Principal Investigator — APHP
Locations (2):
- France (2):
  - Broca Hospital, Paris, Ile de Frane
  - Paul Brousse Hospital, Villejuif, Val De Marne

IPD SHARING:
Plan to Share IPD: No